CLINICAL TRIAL: NCT03888235
Title: Frequency of Sacroiliac Malrotation in Low Back Pain and Correction With a Simple In-home Exercise: A Randomized Study Comparing Those Treated Immediately to Those Waiting One Month for Treatment
Brief Title: Correction of Low Back Pain From Sacroiliac Malrotation With a Simple in Home Exercise
Acronym: SIbackpain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Helene Bertrand, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-01224
Record Dates: First submitted 2019-03-19; First posted 2019-03-25 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Sacroiliac Strain; Low Back Pain
Keywords: Sacroiliac Instability; Sacroiliac Strain; Hypermobility; sacroiliac sprain; tendinopathy
MeSH Terms: conditions — Low Back Pain; Tendinopathy | interventions — Treatment Delay

STUDY DESIGN:
Intervention Model Description: Of all the patients with low back pain, those with sacroiliac malrotation will be randomized to: group 1 an exercise to correct the malrotation, group 2 given a pelvic belt to stabilize the sacroiliac joints, group 3: use of usual treatment and treatment with the belt and exercise one month later. The degree of pain relief and improved function between the first visit and the second visit one month later will be assessed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate corrective exercises (Experimental): At this visit, participants will be examined as described in the protocol and given an exercise to correct their sacroiliac malrotation. They will use this exercise as needed for pain control. They will be reassessed one month later.
  At that time they will be given the pelvic support belt and the concurrent use of both treatments will be assessed at their last visit one month after that.
  Interventions: Procedure: Immediate corrective exercises
- Immediate use of pelvic support belt (Experimental): Participants will be given a pelvic support belt to stabilize their pelvis. They will use this belt for activities likely to precipitate back pain. They will be reassessed one month later.
  At that time they will be given the exercises and the concurrent use of both treatments will be assessed at their last visit one month after that.
  Interventions: Device: Immediate use of pelvic support belt
- Delayed treatment (Active Comparator): These participants will continue using their current therapies to deal with their low back pain for one month prior to being scheduled for a treatment visit. At the treatment visit, one month later they will be given both the exercise and the belt.
  The concurrent use of both treatments will be assessed at their last visit one month after that.
  Interventions: Other: Delayed treatment

INTERVENTIONS:
Procedure: Immediate corrective exercises — The sacroiliac forward flexion test (SIFFT) finds the position of each innominate bone. Subjects learn 1 of 3 exercises. To correct anterior rotation, flex the thigh hard against the ilium, pushing it backwards. To correct posterior rotation, hyperextend the thigh to pull the ilium forward. 1.Genuflect, anterior foot and posterior knee on the floor hands on the floor on either side of the foot, sliding the knee backwards to hyperextend the thigh. 2. Supine, anterior foot on an assistant's sternum, posterior thigh hyperextended. Assistant leans forward, forcing the anterior thigh against the ilium and pushing down on the posterior thigh. 3. For anterior rotation alone: anterior foot on a chair seat, pulling up hard with both hands, leaning back, forcing the thigh against the ilium. Hold position for 2 minutes. Use as needed for pain control. They are reassessed one month later when they receive the pelvic support belt. Both treatments used together will be assessed one month after.
  Other Names: Immediate use of sacroiliac corrective exercises
  Arms: Immediate corrective exercises
Device: Immediate use of pelvic support belt — Participants will be given a pelvic support belt to stabilize their sacroiliac joints. The belt is fitted tightly around the pelvis, over the sacrum and below the anterior superior iliac spines (ASISs) to prevent opening the joint. (The upper part of the innominate bones flares out so pushing them inwards will move the lower part outwards, away from the sacrum, opening the sacroiliac joints, increasing their instability). They will use this belt for activities which have in the past precipitated back pain. They will be reassessed one month later.
  At that time they will be given the exercises to correct their sacroiliac malrotation and the concurrent use of both treatments will be assessed at their last visit one month later.
  Other Names: Serola pelvic support belt
  Arms: Immediate use of pelvic support belt
Other: Delayed treatment — Participants will continue the treatments they are currently using to relieve their low back pain for one month. At their one-month visit, they will be taught how to assess the direction of sacroiliac malrotation and how to do the corrective exercise. They will also be fitted for a pelvic stabilization belt.
  Other Names: One month delay prior to receiving sacroiliac corrective exercises and pelvic support belt
  Arms: Delayed treatment

SUMMARY:
60 participants with low back pain will be examined to determine the direction and extent of sacroiliac malrotation. If malrotation exists, they will be randomized to 3 treatment groups: 1 will be taught how to use their thigh to push the anterior superior iliac spine (ASIS) backwards for an anterior malrotation and their sartorius and rectus femoris to pull their ASIS and anterior inferior iliac spine (AIIS) forward for a posterior malrotation. 2: will be given a pelvic stabilization belt. 3: will return in one month. At the second visit at one month all participants will be treated with both exercise and belt. They will be reassessed at the third visit one month later: the scores for immediate and delayed treatment groups will be compared. Their response to these exercises and/or the pelvic belt will be tested at the first second and third visits, using the brief pain inventory pain, the Oswestry disability scores and the distance between the (posterior superior iliac spine) (PSIS) levels, filled out at every contact. Their satisfaction with previous treatments used will be compared to their satisfaction when using the exercise and belt.

DETAILED DESCRIPTION:
Potential participants with low back pain will answer a questionnaire to eliminate lumbar or hip pathology, ankylosing spondylitis or major leg length discrepancy as cause. If they state they do not have these, they will be given an appointment to be assessed to eliminate the presence of these conditions and to determine if they suffer from sacroiliac malrotation. To this effect, the sacroiliac forward flexion test (SIFFT) will be done: leaning on a counter with their body horizontal to tilt the pelvis forward and lower the sacrum and their legs vertical to push the innominate bones upwards via the hip joints, to expose the posterior superior iliac spines (PSISs). Pressure below the PSISs will be used to assess their inferior limits which will be marked and their levels assessed using a carpenter's level. The distance between the PSIS levels will be recorded. If there is tenderness under the higher PSIS, the ilium is malrotated anteriorly on the sacrum. If the area under the lower PSIS is tender, the ilium is malrotated posteriorly on the sacrum.

Participants are then randomized into three groups: group 1 is taught how to assess the direction of the malrotation, then how to perform the appropriate corrective exercise:

* With the foot of the anteriorly rotated side and the knee on the posteriorly rotated side on the floor, hands on the floor on either side of the foot, the participant leans forward hard to push his anteriorly rotated ilium posteriorly with his thigh and stretches the opposite thigh posteriorly to pull the posteriorly rotated ilium forward.
* Anterior malrotation can also be corrected by placing the foot on the malrotated side on a chair seat, flexing the other knee to touch the seat edge and pulling with both hands up on the seat while leaning back, to drive the thigh against the anterior superior iliac spine (ASIS), thus pushing it backwards.
* If unable to do these, participants can lie supine on the table, thigh on the posterior side extended. On the anterior side the knee is flexed and the foot is on the assistant's sternum as he/she leans forward, pushing the thigh against the ASIS. Downward pressure on the sartorius and rectus femoris just above the knee causes the ASIS and the anterior inferior iliac spine (AIIS) to be pulled on, rotating the ilium anteriorly.

Each position is held for 2 minutes, with up to 2 repetitions as needed. At home, the procedure is repeated as needed for pain relief.

Group 2 are given a pelvic stabilization belt and taught how to apply it: tightly around the pelvis below the anterior superior iliac spines (ASISs), to stabilize the sacroiliac joints as malrotation occurs as a result of pelvic instability. The belt is used for activities known to cause back pain.

Group 3 are instructed to continue their usual treatments and given an appointment to return one month later to receive instruction for the exercise and given the belt At 1 month all are reassessed. Group 1: use and effectiveness of the exercises is recorded and they are given the belt. Group 2: use and effectiveness of the belt is recorded and they are taught how to examine and correct their sacroiliac joints. Group 3: use and satisfaction with their current treatment is recorded. They are then taught the examination and corresponding exercise and given the belt.

At 2 months, when all participants have used both treatments for one month, all are reassessed.

Data collected includes:

at the first visit: Diagnoses associated with low back pain: lumbar spondylosis, hip arthritis, hypermobility, leg length discrepancy.

Conditions associated with sacroiliac malrotation, tendinitis of sacroiliac joint stabilizer muscles and lateral femoral cutaneous neuropathy. Muscle insertions tested include quadratus lumborum, gluteus medius and minimus, piriformis, iliopsoas, biceps femoris, semimembranosus and semitendinosus.

At all visits:

Brief pain inventory pain severity (BPI PS), the Oswestry low-back disability scores (ODI) and the distance in centimetres between the posterior superior iliac spine levels from the SIFFT test (PSISL), at intake, one month and two months visits. Together with the following:

Use of pain medications alcohol and marijuana Use and satisfaction with other treatments for back pain relief (physiotherapy, acupuncture, yoga, core exercises, chiropractor, massage).

Position of the malrotated sacroiliac joint or joints. Distance in centimetres between the levels of the PSISs before and after the corrective exercise. (Visits 2 and 3 for all, visits 1, 2, 3 for group 1) Numeric rating scale pain score after the corrective exercise. Use of and satisfaction with the SI corrective exercise at first visit for group 1 and at the second and third visit for all.

Use of and satisfaction with the pelvic belt at the first visit for group 2 and at the second and third visits for all.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 90
* Participants present with pain in their low back (below the waist) or their buttocks.
* Able to attend all 3 study visits at the participating physician's office.
* Able to attend at least the first two visits with someone willing to assist them in assessing their back and help them with the necessary exercise if need be.
* Willing to perform the corrective exercise and or wear the sacroiliac stabilization belt at home as needed
* Their posterior superior iliac spines (PSISs) are not level on initial examination.
* The long dorsal sacroiliac ligament below at least one of the (PSISs) is tender to palpation on initial examination.

Exclusion Criteria:

* Pain experienced is lumbar in origin
* Pain secondary to hip or other pathology
* PSISs are level at initial examination
* No tenderness to pressure under the PSISs
* Severe pain elsewhere in the body, making the assessment of back pain difficult.
* Presence of ankylosing spondylitis (seen on x-ray, pain worse at night, relieved by exercise, abnormal C reactive protein (CRP) or erythrocyte sedimentation rate (ESR)
* Obvious leg length discrepancy (> 1 ½ cm) when measured umbilicus to medial malleolus.
* Location of PSISs cannot be assessed accurately due to back mice or obesity.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helene Bertrand, Principal Investigator — University of British Columbia Department of family practice
Locations (1):
- Dr. Helene Bertrand Inc., North Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The encrypted de-identified database will be emailed to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will probably be available by December 2020, depending on recruitment.
Access Criteria: Researchers with university affiliation or previous back pain publications or specialists in physical medicine and rehabilitation, pain, neurology, neurosurgery, orthopedic surgery, orthopedic medicine, physiotherapy.

REFERENCES:
- [Background] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Szadek KM, van der Wurff P, van Tulder MW, Zuurmond WW, Perez RS. Diagnostic validity of criteria for sacroiliac joint pain: a systematic review. J Pain. 2009 Apr;10(4):354-68. doi: 10.1016/j.jpain.2008.09.014. Epub 2008 Dec 19. PMID 19101212
- [Result] Potter NA, Rothstein JM. Intertester reliability for selected clinical tests of the sacroiliac joint. Phys Ther. 1985 Nov;65(11):1671-5. doi: 10.1093/ptj/65.11.1671. PMID 2932746
- [Derived] Bertrand H, Reeves KD, Mattu R, Garcia R, Mohammed M, Wiebe E, Cheng AL. Self-Treatment of Chronic Low Back Pain Based on a Rapid and Objective Sacroiliac Asymmetry Test: A Pilot Study. Cureus. 2021 Nov 11;13(11):e19483. doi: 10.7759/cureus.19483. eCollection 2021 Nov. PMID 34912624
- See also: Caitlin R Finley, Derek S Chan, Scott Garrison, et al. What are the most common conditions in primary care? Systematic review, Canadian Family Physician/ Le Médecin De Famille Canadien, 64, November 2018, 832 - 840 — http://www.cfp.ca/content/latest
- See also: Levangie PK , Four clinical tests of sacroiliac joint dysfunction: the association of test results with innominate torsion among patients with and without low back pain. Phys Ther. 1999;79(11):1043. — http://www.physio-pedia.com/Sacroiliac_Joint_Special_Test_Cluster
- See also: Riddle DL, Freburger JK, Evaluation of the presence of sacroiliac joint region dysfunction using a combination of tests: a multicenter intertester reliability study. Phys Ther. 2002;82(8):772. — http://www.lastsite.ca/wp-content/uploads/2016/04/772.full_.pdf
- See also: Description of sacroiliac forward flexion test (SIFFT), the three possible corrective exercises for sacroiliac malrotation, how to apply the pelvic stabilization belt — https://www.youtube.com/watch?v=6phEHENd7jo&t=8s

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Back pain sufferers on a first visit at the doctor's office
Pre-assignment Details: Included were those with evidence of sacroiliac malrotation, excluded were those suffering from sciatic neuropathy, ankylosing spondylitis, hip pathology and leg length discrepancy greater than 3 cm.
Groups:
- Immediate Corrective Exercises: After the sacroiliac forward flexion test (SIFFT) has determined the position of each innominate bone, depending on their ability, subjects are given 1 of 3 exercises to correct their sacroiliac malrotation. All 3 correct anterior malrotation, by flexing the thigh hard against the ilium, pushing it posteriorly. Posterior malrotation, is corrected by hyperextending the thigh, using the sartorius and rectus femoris to pull the ilium anteriorly. These exercises are:
  1. Genuflect, anterior foot and posterior knee on the floor hands on the floor on either side of the foot, sliding the knee backwards to hyperextend the thigh.
  2. In supine position anterior foot on an assistant's sternum, posterior thigh hyperextended. Assistant leans forward, forcing the anterior thigh against the ilium and pushing down on the posterior thigh.
  3. For anterior malrotation alone: anterior foot on a chair seat, pulling up hard with both hands, leaning back, forcing the thigh against the ilium.
  Hold the position for 2 minutes. They will use the exercise as needed for pain control and will be reassessed one month later.
  At that time they will be given the pelvic support belt and the concurrent use of both treatments will be assessed at their last visit one month after that.
- Delayed Treatment: These participants will continue using their current therapies to deal with their low back pain for one month prior to being scheduled for a treatment visit. At the treatment visit, one month later they will be given both the exercise and the belt.
  The concurrent use of both treatments will be assessed at their last visit one month after that.
  Delayed treatment: Participants will continue the treatments they are currently using to relieve their low back pain for one month prior to being treated with the intervention.
Period: Overall Study
Arm/Group | Immediate Corrective Exercises | Immediate Use of Pelvic Support Belt | Delayed Treatment
Started | 21 (1 Participant dropped out after the first visit and was replaced.) | 21 (1 participants dropped out after the first visit and was replaced) | 20
Completed | 20 | 20 | 20
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients with low back pain and sacroiliac malrotation
Groups:
- Delayed Treatment: These participants will continue using their current therapies to deal with their low back pain for one month prior to being scheduled for a treatment visit. At the treatment visit, one month later they will be assessed then given both the exercise and the pelvic stabilization belt to use for one month.
  The concurrent use of both treatments will be assessed at their last visit two months after their initial visit.
- Total: Total of all reporting groups
Arm/Group | Immediate Corrective Exercises | Immediate Use of Pelvic Support Belt | Delayed Treatment | Total
Number analyzed (Participants) | 21 | 21 | 20 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 16 | 51
  >=65 years | 5 | 2 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.14 (15.05) | 51.8 (10.97) | 54.3 (12.94) | 52.03 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 10 | 39
  Male | 6 | 7 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 18 | 14 | 19 | 51
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 1 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 21 | 20 | 62
Sacroiliac Forward Flexion Test (SIFFT) [Mean (Standard Deviation); unit: cm] — Participant stands flexed at the hips, body horizontal, legs vertical. PSISs are located by pressing down with the ulnar side of the thumbs advancing them cephalad towards the PSISs starting on either side of the inter-gluteal cleft. When the PSISs are reached, bony resistance is felt. Ask the participant on which side they feel pain i.e. where the joint is malrotated.
  The examiner then marks the area between his/her thumb and each PSIS. With the participant standing, a horizontal level is placed on the lowest mark and the distance between the level and the highest mark is measured in cm.
  cm | 1.514 (0.688) | 1.286 (0.741) | 1.281 (0.594) | 1.359 (0.676)

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Low-back Pain Disability Questionnaire Score Change Baseline Minus 1 Month: Comparison Immediate Corrective Exercise or Pelvic Stabilization Belt V Delayed: Usual Care
Description: Change in Oswestry low-back disability questionnaire (ODI) score between assessment visit and visit 1 month later. This score is calculated from the sum of the scores in each of 10 sections. Each section is rated 0 for no problem to 5 for complete disability. Section 1, pain intensity, section 2, personal care (washing, dressing etc.), section 3, lifting, section 4, walking, section 5, sitting, section 6, standing, section 7, sleeping, section 8, sex life (if applicable), section 9, social life, section 10, travelling. The score is calculated as: 100 x (sum of the scores in each section / number of sections scored X5). Minimum = 0, maximum = 100. Higher scores mean a worse outcome.
Time Frame: From baseline to 1 month after each participant used their assigned treatment
Population: Participants entering the study all suffered from low back pain from sacroiliac malrotation.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Immediate Corrective Exercises (SIFFTE): After the sacroiliac forward flexion test (SIFFT) has determined the position of each innominate bone, depending on their ability, subjects are given 1 of 3 exercises (SIFFTE) to correct their sacroiliac malrotation. All 3 correct anterior malrotation, by flexing the thigh hard against the ilium, pushing it posteriorly. Posterior malrotation, is corrected by hyperextending the thigh, using the sartorius and rectus femoris to pull the ilium anteriorly. These exercises are:
  1. Genuflect, anterior foot and posterior knee on the floor hands on the floor on either side of the foot, sliding the knee backwards to hyperextend the thigh.
  2. In supine position anterior foot on an assistant's sternum, posterior thigh hyperextended. Assistant leans forward, forcing the anterior thigh against the ilium and pushing down on the posterior thigh.
  3. For anterior malrotation alone: anterior foot on a chair seat, pulling up hard with both hands, leaning back, forcing the thigh against the ilium.
  Hold the position for 2 minutes. They will use the exercise as needed for pain control and will be reassessed one month later.
  At that time they will be given the pelvic support belt and the concurrent use of both treatments will be assessed at their last visit one month after that.
- Immediate Use of Pelvic Support Belt: Participants will be given a pelvic support belt to stabilize their sacroiliac joints. The belt is fitted tightly around the pelvis, over the sacrum and below the anterior superior iliac spines (ASISs) to prevent opening the joint. (The upper part of the innominate bones flares out so pushing them inwards will move the lower part outwards, away from the sacrum, opening the sacroiliac joints, increasing their instability). They will use this belt for activities which have in the past precipitated back pain. They will be reassessed one month later.
  At that time they will be given the exercises to correct their sacroiliac malrotation (SIFFTE) and the concurrent use of both treatments will be assessed at their last visit one month later.
- Delayed Treatment: These participants will continue using their current therapies to deal with their low back pain for one month prior to being scheduled for a treatment visit. At the treatment visit, one month later they will be given both the corrective exercise (SIFFTE) and the pelvic support belt.
  The concurrent use of both treatments, the corrective exercise (SIFFTE) and the pelvic support belt will be assessed at their last visit one month after that.
Arm/Group | Immediate Corrective Exercises (SIFFTE) | Immediate Use of Pelvic Support Belt | Delayed Treatment
Number analyzed (Participants) | 21 | 21 | 20
score on a scale | 8 [0 to 19] | 2 [-4 to 9] | -2.4 [-6 to 6]
Statistical Analysis 1: Comparison: Immediate Corrective Exercises (SIFFTE) vs Immediate Use of Pelvic Support Belt vs Delayed Treatment; The null hypothesis assumes that after one month, there is no difference in Oswestry low back pain and disability score improvement between the three treatment groups; Test type: Superiority; p = 0.003, Kruskal-Wallis
Statistical Analysis 2: Comparison: Immediate Corrective Exercises (SIFFTE) vs Delayed Treatment; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney) — SI Exercise versus usual care. Bonferroni alpha correction p< 0.0167
Statistical Analysis 3: Comparison: Immediate Use of Pelvic Support Belt vs Delayed Treatment; Null hypothesis: there is no difference in Oswestry low back pain and disability score between those using a pelvic support belt and those using usual treatment; Test type: Superiority; p = 0.314, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Oswestry Low-Back Pain Disability Questionnaire Score Change Baseline Minus 2 Month Score, After One Month Of Using Corrective Exercise + Pelvic Stabilization Belt
Description: Change in Oswestry low-back disability questionnaire (ODI) score between assessment visit and visit 2 months later after using the corrective exercise + the pelvic stabilization belt for one month. =(ODI at assessment - ODI at 2 months). The ODI score is calculated from the sum of the scores in each of 10 sections. Each section is rated 0 for no problem to 5 for complete disability. Section 1, pain intensity, section 2, personal care (washing, dressing etc.), section 3, lifting, section 4, walking, section 5, sitting, section 6, standing, section 7, sleeping, section 8, sex life (if applicable), section 9, social life, section 10, travelling. The score is calculated as: 100 x (sum of the scores in each section / number of sections scored). Minimum = 0, maximum = 100. Higher scores mean greater disability, a worse outcome. The greater the change, the better the outcome.
Time Frame: Two months: from baseline visit to last visit two months later when all participants have used both the pelvic stabilization belt and the corrective exercise for one month
Population: All participants, Oswestry low-back pain disability questionnaire score change: baseline minus the score two months later after one month of use of corrective exercises and sacroiliac stabilization belt.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Baseline Oswestry Disability Index (ODI) Score: All participants received the Oswestry Disability Index ODI questionnaire on being admitted in the study. The ODI score is calculated from the sum of the scores in each of 10 sections. Each section is rated 0 for no problem to 5 for complete disability. Section 1, pain intensity, section 2, personal care (washing, dressing etc.), section 3, lifting, section 4, walking, section 5, sitting, section 6, standing, section 7, sleeping, section 8, sex life (if applicable), section 9, social life, section 10, travelling. The score is calculated as: 100 x (sum of the scores in each section / number of sections scored X5). Minimum = 0, maximum = 100. Higher scores mean a worse outcome.
- ODI After Immediate Corrective Exercises + Sacroiliac Stabilization Belt Used For One Month: All participants get the sacroiliac forward flexion test (SIFFT): standing, trunk forward flexed the posterior superior iliac spine (PSIS) levels are found and measured. A higher painful PSIS has anterior, a lower one has posterior malrotation. They are given the appropriate exercise to correct their sacroiliac malrotation. Anterior rotation is corrected with the flexed thigh pushing hard on the anterior superior iliac spine to force it posteriorly. Posterior rotation is corrected by hyperextending the thigh, using the sartorius and the rectus femoris to pull the ilium anteriorly. 3 techniques: - genuflection, anterior side foot and posterior side knee on the floor, hands on either side of the foot, knee stretched backwards, - anterior side foot on chair, pull up on chair to force the thigh against the ilium, - in dorsal decubitus assistant with anterior side foot on their sternum leans forward to push the thigh against ilium and pushes down on extended posterior side thigh to overstretch it. All these are held for 2 minutes. They are then fitted with a sacroiliac stabilization belt to wear as needed for back pain producing activities. They are reassessed using the Oswestry disability Index score (ODI) one month later at their two month visit.
Arm/Group | Baseline Oswestry Disability Index (ODI) Score | ODI After Immediate Corrective Exercises + Sacroiliac Stabilization Belt Used For One Month
Number analyzed (Participants) | 62 | 62
score on a scale | 36 [26 to 46] | 23.11 [14 to 38]
Statistical Analysis 1: Comparison: Baseline Oswestry Disability Index (ODI) Score; Oswestry low back pain and disability (ODI) score change over two months for all participants. This compares the score at initial visit and the score 2 months later after all participants have been using the corrective exercise and sacroiliac stabilization belt for one month. =(ODI time 0 - ODI 2 months). The greater the difference, the better the recovery of back function; Test type: Superiority; p < 0.001, Kruskal-Wallis

3. Secondary Outcome: Brief Pain Inventory Score Change Over One Month. Baseline Score Minus 1 Month Score. Comparison: Immediate Corrective Exercise or Pelvic Stabilization Belt V Delayed: Usual Care
Description: Change in BPI pain score between baseline assessment visit and visit one month later: on a scale of 0 (no pain) to 10 (worst imaginable pain) pain in the last 24 hours:
  • on average • at its worst • at its best • right now. Average of these values. Minimum value, 0, maximum value, 10. Higher scores mean a worse outcome. A higher change between the initial visit and the one month visit means a better outcome.
Time Frame: 1 month after initial visit (baseline BPI pain score minus one-month BPI pain score) with each group using their assigned treatment
Population: People with low back pain and malrotated sacroiliac joints.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Immediate Corrective Exercises | Immediate Use of Pelvic Support Belt | Delayed Treatment
Number analyzed (Participants) | 21 | 21 | 20
score on a scale | 1.25 [0.25 to 2.25] | 1 [0.75 to 2.875] | 0.25 [-.75 to 1.5]
Statistical Analysis 1: Comparison: Immediate Corrective Exercises vs Immediate Use of Pelvic Support Belt vs Delayed Treatment; The null hypothesis assumes that after one month, there is no difference in brief pain inventory score improvement between the three treatment groups; Test type: Superiority; p = 0.17, Kruskal-Wallis
Statistical Analysis 2: Comparison: Immediate Corrective Exercises vs Delayed Treatment; The brief pain inventory score at the one month visit, is used to compare the pain levels of those having done one month of corrective exercises to those who continued with conventional treatments for their low back pain; Test type: Superiority; p = 0.089, Wilcoxon (Mann-Whitney) — Bonferroni alpha correction of p<0.0167
Statistical Analysis 3: Comparison: Immediate Use of Pelvic Support Belt vs Delayed Treatment; The brief pain inventory score is used to compare those using a pelvic support belt for one month and those with delayed treatment; Test type: Superiority; p = 0.092, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Brief Pain Inventory (BPI) Pain Score Change Over Two Months Comparison: Baseline (BPI) Pain Score Minus 2 Month (BPI) Pain Score, After One Month Of Using Corrective Exercise + Pelvic Stabilization Belt
Description: Change in BPI pain score between baseline visit and visit minus BPI pain score two months later after one month of using corrective exercise + pelvic stabilization belt On a scale of 0 (no pain) to 10 (worst imaginable pain) pain in the last 24 hours: • on average • at its worst • at its best • right now. Average of these values. Minimum value, 0, maximum value, 10. Higher scores mean a worse outcome. A higher change between the initial visit and the later visit means a better outcome.
Time Frame: 2 months after baseline visit when all groups have used both the pelvic stabilization belt and the corrective exercise for one month
Population: People with low back pain and malrotated sacroiliac joints.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Initial Brief Pain Inventory (BPI) Pain Score: At their initial visit, all participants fill out the brief pain inventory (BPI) pain score: on a scale of 0 (no pain) to 10 (worst imaginable pain) pain in the last 24 hours:
  • on average • at its worst • at its best • right now. Average of these values. Minimum value, 0, maximum value, 10. Higher scores mean a worse outcome. A higher change between the initial visit and the one month visit means a better outcome.
- Corrective Exercises (SIFFTE) Plus Sacroiliac Belt Use For One Month: Effect on (BPI) Pain Score: All participants fill out the brief pain inventory pain score (BPI) then get the sacroiliac forward flexion test (SIFFT): standing, trunk forward flexed the posterior superior iliac spine levels (PSISL) are found and measured. A higher painful PSIS has anterior, a lower one has posterior malrotation. They are given the appropriate exercise (PSISE) to correct their sacroiliac malrotation. Anterior rotation is corrected with the flexed thigh pushing hard on the anterior superior iliac spine to force it posteriorly. Posterior rotation is corrected by hyperextending the thigh, using the sartorius and the rectus femoris to pull the ilium anteriorly. 3 techniques: - genuflection, anterior side foot and posterior side knee on the floor, hands on either side of the foot, knee stretched backwards, - anterior side foot on chair, pull up on chair to force the thigh against the ilium, - in dorsal decubitus assistant with anterior side foot on their sternum leans forward to push the thigh against ilium and pushes down on extended posterior side thigh to overstretch it. All these are held for 2 minutes. They are then fitted with a sacroiliac stabilization belt to wear as needed for back pain producing activities. They are reassessed one month later at their two month visit once again using the BPI pain score.
Arm/Group | Initial Brief Pain Inventory (BPI) Pain Score | Corrective Exercises (SIFFTE) Plus Sacroiliac Belt Use For One Month: Effect on (BPI) Pain Score
Number analyzed (Participants) | 62 | 62
score on a scale | 5.88 [4.5 to 7.25] | 3.5 [1.75 to 5.25]
Statistical Analysis 1: Comparison: Initial Brief Pain Inventory (BPI) Pain Score vs Corrective Exercises (SIFFTE) Plus Sacroiliac Belt Use For One Month: Effect on (BPI) Pain Score; All participants are assessed as a single group as they receive the same two treatments for one month. Brief pain inventory (BPI) score change over two months for all participants. This compares BPI score at baseline visit and BPI score 2 months later, after all participants have been using the corrective exercise and sacroiliac stabilization belt for one month. The score is between 0 and 10. The higher the change in score the greater the pain relief; Test type: Superiority; p < 0.001, Kruskal-Wallis

5. Secondary Outcome: Distance Between The Posterior Superior Iliac Spine Levels (PSISL) Using The Sacroiliac Forward Flexion (SIFFT) Test Comparing Corrective Exercise, Pelvic Belt, Conventional Treatment: Baseline Value Minus 1 Month Value..
Description: Difference in distance in centimetres between the levels of the higher & the lower posterior superior iliac spines as measured using a carpenter's level between the value found on admission and that found one month later (PSISL). The minimum is 0 cm, the maximum is 3.5 cm. Higher scores mean a worse outcome. The greater difference when the distance is calculated between admission and one or two months later means a better outcome.
Time Frame: One month comparing the different treatments at baseline and one month later.
Population: People with back pain and malrotated sacroiliac joints
Measure: Median (Inter-Quartile Range); unit: cm
Groups:
- Immediate Corrective Exercises (SIFFTE): The sacroiliac forward flexion test (SIFFT) will determine the level of each posterior superior iliac spine (PSISL). The distance in centimetres between the levels of the PSISs will be recorded. Depending on their ability, subjects are given 1 of 3 exercises to correct their sacroiliac malrotation. All 3 correct anterior malrotation by flexing the thigh hard against the ilium, pushing it posteriorly. Posterior malrotation, is corrected by hyperextending the thigh, using the sartorius and rectus femoris to pull the ilium anteriorly. These exercises are:
  1. Genuflect, anterior foot and posterior knee on the floor hands on the floor on either side of the foot, sliding the knee backwards to hyperextend the thigh.
  2. In supine position anterior foot on an assistant's sternum, posterior thigh hyperextended. Assistant leans forward, forcing the anterior thigh against the ilium and pushing down on the posterior thigh.
  3. For anterior malrotation alone: anterior foot on a chair seat, pulling up hard with both hands, leaning back, forcing the thigh against the ilium.
  Hold the position for 2 minutes. They will use the exercise as needed for pain control and will be reassessed with the PSISL one month later.
  At that time they will be given the pelvic support belt. The concurrent use of both treatments will be assessed at their last visit one month later using the PSISL.
- Immediate Use of Pelvic Support Belt: The sacroiliac forward flexion test (SIFFT) will determine the level of each posterior superior iliac spine (PSISL). The distance in centimetres between the levels of the PSISs will be recorded. Following this, participants will be given a pelvic support belt to stabilize their sacroiliac joints. The belt is fitted tightly around the pelvis, over the sacrum and below the anterior superior iliac spines (ASISs) to prevent opening the joint. (The upper part of the innominate bones flares out so pushing them inwards will move the lower part outwards, away from the sacrum, opening the sacroiliac joints, increasing their instability). They will use this belt for activities which have in the past precipitated back pain. They will be reassessed one month later with the PSISL.
  At that time they will be given the exercises to correct their sacroiliac malrotation and the concurrent use of both treatments will be assessed with the PSISL at their last visit one month later.
- Delayed Treatment: The sacroiliac forward flexion test (SIFFT) will determine the level of each posterior superior iliac spine (PSISL). The distance in centimetres between the levels of the PSISs will be recorded. These participants will continue using their current therapies to deal with their low back pain for one month prior to being scheduled for a treatment visit. At the treatment visit, one month later they will be given both the corrective exercise (SIFFTE) and the pelvic support belt after their PSISL has been recorded.
  The concurrent use of both treatments will be assessed using the PSISL at their last visit one month after that.
  Delayed treatment: Participants will continue the treatments they are currently using to relieve their low back pain for one month prior to being treated with the intervention.
Arm/Group | Immediate Corrective Exercises (SIFFTE) | Immediate Use of Pelvic Support Belt | Delayed Treatment
Number analyzed (Participants) | 21 | 21 | 20
cm | 1.375 [0.25 to 2.25] | 1.125 [-.125 to 2.875] | 0.25 [-.875 to 1.875]
Statistical Analysis 1: Comparison: Immediate Corrective Exercises (SIFFTE) vs Immediate Use of Pelvic Support Belt vs Delayed Treatment; The null hypothesis assumes there is no improvement after one month in posterior superior iliac spine levels (PSISL) measured using the sacroiliac forward flexion test (SIFFT) between the three treatment groups; Test type: Superiority; p = 0.016, Kruskal-Wallis — The Bonferroni alpha correction is used p<0.0167
Statistical Analysis 2: Comparison: Immediate Corrective Exercises (SIFFTE) vs Delayed Treatment; The null hypothesis is that there is no difference in the distance between the posterior sacroiliac spine levels (PSISL) between those who use their usual low back pain treatments and those who are given the corrective exercises (SIFFTE) and use them as needed for one month; Test type: Superiority; p = 0.009, Wilcoxon (Mann-Whitney) — The Bonferroni alpha correction is used p<0.0167
Statistical Analysis 3: Comparison: Immediate Use of Pelvic Support Belt vs Delayed Treatment; The null hypothesis is that that using a pelvic support belt will not help correct sacroiliac joint asymmetry as measured using the distance between the posterior superior iliac spine levels (PSISL), baseline and one month later better than conventional treatment for low back pain; Test type: Superiority; p = 0.034, Wilcoxon (Mann-Whitney) — Bonferroni correction p< 0.0167

6. Secondary Outcome: Distance Between The Posterior Superior Iliac Spine Levels (PSISL) Using The Sacroiliac Forward Flexion (SIFFT) Test, Baseline Minus One Month After Using Corrective Exercise (SIFFTE) + Pelvic Stabilization Belt.
Description: The distance between the levels (determined using a carpenter's level) of the higher & the lower posterior superior iliac spines (PSISL) was measured in centimetres. The outcome measure is the difference between the value found on admission and that (PSISL) value found two months later after all participants have use the corrective exercises (SIFFT E) and the sacroiliac stabilizer belt for one month. The minimum is 0 cm, the maximum is 3.5 cm. On admission, higher scores mean a worse outcome. The greater difference when the distance is calculated between admission and two months later means a better outcome.
Time Frame: 2 months: comparing baseline values and values after all participants have used the corrective exercise and the sacroiliac stabilization belt for one month.
Population: People with back pain and malrotated sacroiliac joints. Corona virus pandemic prevented 28 participants from returning for a final examination.
Measure: Median (Inter-Quartile Range); unit: cm
Groups:
- Baseline Recording of the Distance Between Posterior Superior Iliac Spine Levels (PSISL): On admission into the study, all participants get the sacroiliac forward flexion test (SIFFT): standing, trunk forward flexed the posterior superior iliac spine (PSIS) levels are found and the distance between them is measured in centimetres.
- Immediate Corrective Exercises And Use Of Pelvic Stabilization Belt For One Month: At their second visit, one month after the baseline visit, all participants get the sacroiliac forward flexion test (SIFFT): standing, trunk forward flexed the posterior superior iliac spine (PSIS) levels are found and the distance between these is recorded (PSISL). A higher painful PSIS has anterior, a lower one has posterior malrotation. They are given the appropriate exercise to correct their sacroiliac malrotation. Anterior rotation is corrected with the flexed thigh pushing hard on the anterior superior iliac spine to force it posteriorly. Posterior rotation is corrected by hyperextending the thigh, using the sartorius and the rectus femoris to pull the ilium anteriorly. 3 techniques: - genuflection, anterior side foot and posterior side knee on the floor, hands on either side of the foot, knee stretched backwards, - anterior side foot on chair, pull up on chair to force the thigh against the ilium, - in dorsal decubitus assistant with anterior side foot on their sternum leans forward to push the thigh against ilium and pushes down on extended posterior side thigh to overstretch it. All these are held for 2 minutes. They are then fitted with a sacroiliac stabilization belt to wear as needed for back pain producing activities. They are reassessed (PSISL) one month later at their two month visit.
Arm/Group | Baseline Recording of the Distance Between Posterior Superior Iliac Spine Levels (PSISL) | Immediate Corrective Exercises And Use Of Pelvic Stabilization Belt For One Month
Number analyzed (Participants) | 33 | 33
cm | 1.2 [1 to 1.9] | 0.3 [0 to 1]
Statistical Analysis 1: Comparison: Baseline Recording of the Distance Between Posterior Superior Iliac Spine Levels (PSISL) vs Immediate Corrective Exercises And Use Of Pelvic Stabilization Belt For One Month; Since all participants have received the same 2 treatment for one month, we will treat them as a single group. We will measure the distance between their posterior superior iliac spine levels (PSISL) when they enter the study and two months later after they have used the corrective exercise and the sacroiliac belt for one month. Corona prevented some participants from returning for examination, which this test requires. Only 11 participants were present in each group: 33 participants tested; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline Recording of the Distance Between Posterior Superior Iliac Spine Levels (PSISL) vs Immediate Corrective Exercises And Use Of Pelvic Stabilization Belt For One Month; Test type: Superiority; p < 0.001, Kruskal-Wallis

7. Post Hoc Outcome: Satisfaction Level With Physiotherapy Baseline Compared To Satisfaction Level With The Corrective Exercise (SIFFTE) Plus The Pelvic Support Belt Used For One Month
Description: At baseline, participants answered the satisfaction questionnaire: "on a scale of 0 - 3 where 0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always, how satisfied were you with physiotherapy?" Two months later, after using the corrective exercise (SIFFTE) and the pelvic support belt for one month they were asked the same satisfaction questions for the corrective exercise (SIFFTE) and the pelvic support belt, following which they were asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. The minimum value was 0, the maximum value was 3. Higher scores mean a better outcome.
Time Frame: 2 months
Population: Participants in the study who had received physiotherapy treatments prior to entering the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfaction With Physiotherapy: Participants joining the study having previously received physiotherapy treatments. On joining the study they rated their satisfaction with this treatment from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied).
- Satisfaction With Corrective Exercise (SIFFTE) and Pelvic Belt: After the sacroiliac forward flexion test (SIFFT) determined the position of each innominate bone, depending on their ability, subjects were given 1 of 3 exercises (SIFFTE) to correct their sacroiliac malrotation. All 3 correct anterior malrotation, by flexing the thigh hard against the ilium, pushing it posteriorly. Posterior malrotation, is corrected by hyperextending the thigh, using the sartorius and rectus femoris to pull the ilium anteriorly. One of 3 different exercises was used depending on the participants' ability to perform them.
  The position is held for 2 minutes. They used the exercise as needed for pain control.
  Participants were also given a pelvic support belt to stabilize their sacroiliac joints. The belt is fitted tightly around the pelvis, over the sacrum and below the anterior superior iliac spines (ASISs) to prevent opening the joint. (The upper part of the innominate bones flares out so pushing them inwards will move the lower part outwards, away from the sacrum, opening the sacroiliac joints, increasing their instability). They used this belt for activities which had in the past precipitated back pain.
  They were reassessed one month later. At that time, they were asked how satisfied they were with each treatment on a scale from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied) and which treatment they preferred, exercise, belt, both or neither. The score for the preferred therapy was recorded.
Arm/Group | Satisfaction With Physiotherapy | Satisfaction With Corrective Exercise (SIFFTE) and Pelvic Belt
Number analyzed (Participants) | 47 | 47
score on a scale | 1.02 (0.89) | 2.32 (0.81)
Statistical Analysis 1: Comparison: Satisfaction With Physiotherapy vs Satisfaction With Corrective Exercise (SIFFTE) and Pelvic Belt; the null hypothesis is that all participants were as satisfied with the physiotherapy as they were with using the corrective exercises and the pelvic stabilization belt; Test type: Superiority; p < 0.00001, t-test, 2 sided

8. Post Hoc Outcome: Satisfaction Level With Acupuncture Baseline Compared To Satisfaction Level With The Corrective Exercise (SIFFTE) Plus The Pelvic Support Belt Used For One Month
Description: At baseline, participants answered the satisfaction questionnaire: "on a scale of 0 - 3 where 0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always, how satisfied were you with acupuncture?" Two months later, after using the corrective exercise (SIFFTE) and the pelvic support belt for one month they were asked the same satisfaction questions for the corrective exercise (SIFFTE) and the pelvic support belt, following which they were asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. The minimum value was 0, the maximum value was 3. Higher scores mean a better outcome.
Time Frame: 2 months
Population: All participants who entered the study having previously received acupuncture
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfaction With Acupuncture: Participants joining the study having previously received acupuncture treatments. On joining the study they rated their satisfaction with this treatment from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied).
- Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt: After the sacroiliac forward flexion test (SIFFT) determined the position of each innominate bone, depending on their ability, subjects were given 1 of 3 exercises (SIFFTE) to correct their sacroiliac malrotation. All 3 correct anterior malrotation, by flexing the thigh hard against the ilium, pushing it posteriorly. Posterior malrotation, is corrected by hyperextending the thigh, using the sartorius and rectus femoris to pull the ilium anteriorly. One of 3 different exercises was used depending on the participants' ability to perform them.
  The position is held for 2 minutes. They used the exercise as needed for pain control.
  Participants were also given a pelvic support belt to stabilize their sacroiliac joints. The belt is fitted tightly around the pelvis, over the sacrum and below the anterior superior iliac spines (ASISs) to prevent opening the joint. (The upper part of the innominate bones flares out so pushing them inwards will move the lower part outwards, away from the sacrum, opening the sacroiliac joints, increasing their instability). They used this belt for activities which had in the past precipitated back pain.
  They were reassessed one month later. At that time, they were asked how satisfied they were with each treatment on a scale from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied) and which treatment they preferred, exercise, belt, both or neither. The score for the preferred therapy was recorded.
Arm/Group | Satisfaction With Acupuncture | Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt
Number analyzed (Participants) | 34 | 34
score on a scale | 0.97 (0.71) | 2.41 (0.7)
Statistical Analysis 1: Comparison: Satisfaction With Acupuncture vs Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt; the null hypothesis is that all participants were as satisfied with the acupuncture as they were with using the corrective exercises and the pelvic stabilization belt; Test type: Superiority; p < 0.00001, t-test, 2 sided

9. Post Hoc Outcome: Satisfaction Level With Yoga Baseline Compared to Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt Used for One Month
Description: At baseline, participants answered the satisfaction questionnaire: "on a scale of 0 - 3 where 0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always, how satisfied were you with doing yoga?" Two months later, after using the corrective exercise (SIFFTE) and the pelvic support belt for one month they were asked the same satisfaction questions for the corrective exercise (SIFFTE) and the pelvic support belt, following which they were asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. The minimum value was 0, the maximum value was 3. Higher scores mean a better outcome.
Time Frame: 2 months
Population: All participants who entered the study having previously participated in yoga exercises
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfaction With Yoga: Participants joining the study having previously participated in yoga exercises. On joining the study they rated their satisfaction with this treatment from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied).
- Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Beltbelt: As part of this study they were given the corrective exercise for their malrotated sacroiliac joint as well as the pelvic stabilization belt and used these for one month. After this month, two months after joining the study, they rated their satisfaction with the corrective exercise (SIFFTE) from 0 - 3 and with the pelvic stabilization belt from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied). They were then asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used.
Arm/Group | Satisfaction With Yoga | Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Beltbelt
Number analyzed (Participants) | 27 | 27
score on a scale | 0.92 (0.83) | 2.37 (0.84)
Statistical Analysis 1: Comparison: Satisfaction With Yoga vs Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Beltbelt; The null hypothesis is that all participants were as satisfied with the yoga exercises as they were with using the corrective exercises and the pelvic stabilization belt; Test type: Superiority; p < 0.00001, t-test, 2 sided

10. Post Hoc Outcome: Satisfaction Level With Core Exercises Baseline Compared to Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt Used for One Month
Description: At baseline, participants answered the satisfaction questionnaire: "on a scale of 0 - 3 where 0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always, how satisfied were you with doing core exercises?" Two months later, after using the corrective exercise (SIFFTE) and the pelvic support belt for one month they were asked the same satisfaction questions for the corrective exercise (SIFFTE) and the pelvic support belt, following which they were asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. The minimum value was 0, the maximum value was 3. Higher scores mean a better outcome.
Time Frame: 2 months
Population: All participants who entered the study having previously performed core exercises
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfaction With Core Exercises: Participants joining the study having previously participated in core exercises. On joining the study they rated their satisfaction with this treatment from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied).
- Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt: As part of this study they were given the corrective exercise (SIFFTE) for their malrotated sacroiliac joint as well as the pelvic stabilization belt and used these for one month. After this month, two months after joining the study, they rated their satisfaction with the corrective exercise (SIFFTE) from 0 - 3 and with the pelvic stabilization belt from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied). They were then asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. Wow that's impressive her be and I have done have been 10,802 and 41
Arm/Group | Satisfaction With Core Exercises | Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt
Number analyzed (Participants) | 38 | 38
score on a scale | 1.08 (0.78) | 2.21 (0.81)
Statistical Analysis 1: Comparison: Satisfaction With Core Exercises vs Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt; the null hypothesis is that all participants were as satisfied with the core exercises as they were with using the corrective exercise and the pelvic stabilization belt; Test type: Superiority; p < 0.00001, t-test, 2 sided

11. Post Hoc Outcome: Satisfaction Level With Chiropractic Manipulation Baseline Compared to Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt Used for One Month
Description: At baseline, participants answered the satisfaction questionnaire: "on a scale of 0 - 3 where 0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always, how satisfied were you with the treatments you received from your chiropractor?" Two months later, after using the corrective exercise (SIFFTE) and the pelvic support belt for one month they were asked the same satisfaction questions for the corrective exercise (SIFFTE) and the pelvic support belt, following which they were asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. The minimum value was 0, the maximum value was 3. Higher scores mean a better outcome.
Time Frame: 2 months
Population: All participants who entered the study having previously received treatment by a chiropractor
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfaction With the Treatments Received From a Chiropractor: Participants joining the study having previously received chiropractic treatments. On joining the study they rated their satisfaction with this treatment from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied).
- Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt: As part of this study they were given the corrective exercise (SIFFTE) for their malrotated sacroiliac joint as well as the pelvic stabilization belt and used these for one month. After this month, two months after joining the study, they rated their satisfaction with the corrective exercise (SIFFTE) from 0 - 3 and with the pelvic stabilization belt from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied). They were then asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used.
Arm/Group | Satisfaction With the Treatments Received From a Chiropractor | Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt
Number analyzed (Participants) | 42 | 42
score on a scale | 1 (0.91) | 2.28 (0.83)
Statistical Analysis 1: Comparison: Satisfaction With the Treatments Received From a Chiropractor vs Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt; the null hypothesis is that all participants were as satisfied with treatments by a chiropractor as they were with using the corrective exercise and the pelvic stabilization belt; Test type: Superiority; p < 0.00001, t-test, 2 sided

12. Post Hoc Outcome: Satisfaction Level With Massage Therapy Baseline Compared to Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt Used For One Month
Description: At baseline, participants answered the satisfaction questionnaire: "on a scale of 0 - 3 where 0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always, how satisfied were you with massage therapy?" Two months later, after using the corrective exercise (SIFFTE) and the pelvic support belt for one month they were asked the same satisfaction questions for the corrective exercise (SIFFTE) and the pelvic support belt, following which they were asked whether they preferred the exercise, the belt, both or neither. If they chose the exercise, the satisfaction score for the exercise was used, if they chose the belt the satisfaction score for the belt was used, if they chose both the higher satisfaction score was used, if they chose neither the lower satisfaction score was used. The minimum value was 0, the maximum value was 3. Higher scores mean a better outcome.
Time Frame: 2 months
Population: All participants who entered the study having previously received massage therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Satisfaction With Massage Therapy: Participants joining the study having previously received massage therapy. On joining the study they rated their satisfaction with this treatment from 0 - 3. (0 = not at all, 1 = sometimes, 2 = most of the time, 3 = always satisfied).
Arm/Group | Satisfaction With Massage Therapy | Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt
Number analyzed (Participants) | 42 | 42
score on a scale | 1.19 (0.86) | 2.36 (0.73)
Statistical Analysis 1: Comparison: Satisfaction With Massage Therapy vs Satisfaction With Corrective Exercises (SIFFTE) and Pelvic Support Belt; The null hypothesis is that all participants were as satisfied with massage therapy as they were with using the corrective exercise and the pelvic stabilization belt; Test type: Superiority; p < 0.00001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The timeframe was two months from the time of the baseline assessment and assignment to a treatment group to 2 months later after all participants had used both the corrective exercises (SIFFTE) and the pelvic stabilization belt for one month.
Arm/Group | Immediate Corrective Exercises | Immediate Use of Pelvic Support Belt | Delayed Treatment
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 6/21 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Corrective Exercises (N=21) | Immediate Use of Pelvic Support Belt (N=21) | Delayed Treatment (N=20)
rash, skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) — The foam rubber backing of the pelvic stabilization belt directly against the skin caused irritation.
Unspecified pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) — 1 Uncomfortable at night, 1 feelings of restricted blood flow, 1 increased pain, 1 sometimes caused pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03888235/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03888235/ICF_002.pdf